CLINICAL TRIAL: NCT02165293
Title: A Single Center Study to Evaluate the Penetration of RO7033877 Into the Lung in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: NP29332
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Bronchoscopy

ARMS (1):
- RO7033877 (Experimental)
  Interventions: Drug: RO7033877 + Bronchoscopy

INTERVENTIONS:
Drug: RO7033877 + Bronchoscopy — Days 1, 2, and 3: 2.5 mg/kg RO7033877 infused IV over 2 hours, every 8 hours for a total of 7 doses; BAL procedure on Day 3.

SUMMARY:
This single-center, open-label study will investigate RO7033877 concentrations in plasma and in various lung compartments, including epithelial lining fluid (ELF), and alveolar macrophages (AM) in healthy volunteers after multiple intravenous (IV) administration. Bronchoscopy will be performed after the start of the last infusion on Day 3 at different timepoints. Blood, urine and brochoalveolar lavage samples will be collected to determine RO7033877 concentrations. The anticipated time on study treatment is 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers, 18 to 55 years of age, inclusive. A female participant is eligible to participate if she is of non-childbearing potential defined as postmenopausal or surgically sterile
* Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, serology and urinalysis
* Body mass index (BMI) between 18 and 30 kg/m2 inclusive
* Nonsmokers
* Healthy male volunteers with female partners of childbearing potential must use adequate contraception methods

Exclusion Criteria:

* Evidence of active chronic disease
* Regular consumption of drugs of abuse
* Infection with human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV)
* History of clinically significant hypersensitivity or allergic drug reactions
* Clinically significant abnormalities (e.g. cardiovascular, laboratory values)
* Abnormal blood pressure or vital signs
* Contraindications to bronchoalveolar lavage (BAL)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Multiple-dose pharmacokinetics of RO7033877 for plasma, epithelial lining fluid (ELF), and alveolar macrophage (AM): Cmax and AUC | 5 days (in-clinic period)
ELF and AM/Plasma Ratios of Cmax and AUC | 5 days (in-clinic period)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 12 days
Changes in clinical laboratory safety tests, vital signs, and ECGs | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Phoenix, Arizona, United States